CLINICAL TRIAL: NCT07381569
Title: A Clinical Study on the Safety and Efficacy of Estradiol-Loaded Silicone Rubber Intrauterine Stent System for Promoting Endometrial Repair After Induced Abortion
Brief Title: To Study the Safety and Efficacy of A Novel Intrauterine Estrogen-Releasing System in Induced Abortion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K8309
Record Dates: First submitted 2025-11-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Abortion, Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estradiol-Loaded Silicone Rubber Intrauterine Stent System (Experimental)
  Interventions: Device: Estradiol-Loaded Silicone Rubber Intrauterine Stent System
- No-Drug-Loaded Silicone Rubber Intrauterine Stent System (Sham Comparator)
  Interventions: Device: No-Drug-Loaded Silicone Rubber Intrauterine Stent System

INTERVENTIONS:
Device: Estradiol-Loaded Silicone Rubber Intrauterine Stent System — After abortion, an estradiol-loaded silicone rubber intrauterine stent system was placed for 21+2 days, and oral anti-infective medication was administered for 3 days postoperatively.
  Arms: Estradiol-Loaded Silicone Rubber Intrauterine Stent System
Device: No-Drug-Loaded Silicone Rubber Intrauterine Stent System — After abortion, a no-drug-loaded silicone rubber intrauterine stent system was placed for 21+2 days, and oral anti-infective medication was administered for 3 days postoperatively.
  Arms: No-Drug-Loaded Silicone Rubber Intrauterine Stent System

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of the estradiol-loaded silicone rubber intrauterine stent system for promoting endometrial repair after artificial abortion. The main research questions it aims to answer are:

1. Can the estradiol-loaded silicone rubber intrauterine stent system increase the endometrial thickness at 21+2 days after the procedure?
2. What adverse events or safety issues occur in participants when using this product? Researchers will compare the estradiol-loaded silicone rubber intrauterine stent system with a non-drug-loaded silicone intrauterine stent to determine whether the drug-eluting stent offers advantages in promoting endometrial repair.

Participants will:

1. Undergo placement of either the estradiol-eluting stent or the non-drug stent immediately after artificial abortion, with the stent retained for 21+2 days
2. Attend scheduled follow-up visits at 21+2 days, after the first menstruation, and at 90 days post-procedure.
3. Undergo ultrasound examinations to measure endometrial thickness, and record vaginal bleeding duration, blood loss volume, time to first menstruation, and any adverse events

ELIGIBILITY:
Inclusion Criteria

1. Female patients aged 18-40 years；
2. Menstrual cycle was 21-35 days within the six months before enrollment；
3. BMI between 18.5-28 kg/m²；
4. Voluntary termination of pregnancy, history of ≥2 abortions or missed abortion, and confirmed gestational age ≤10 weeks；
5. Willing to participate, able to attend regular follow-ups, and sign the informed consent form.

Exclusion Criteria

1. Known allergy or contraindication to silicone rubber or estrogen；
2. History of hysteroscopically confirmed uterine adhesions or diagnosed thin endometrium；
3. Uterine malformation, uterine fibroids compressing the uterine cavity, or other causes of abnormal uterine cavity shape；
4. Participants requesting IUD placement, oral contraceptives, or subcutaneous implantation after surgery；
5. Patients with mental or cognitive impairment, unable to cooperate with the treatment process；
6. Patients considered by the investigator to have potential risks or factors making them unsuitable for inclusion.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | at 21 + 2 Days Postoperatively
  Measured via transvaginal ultrasound (unit: mm). The measurement is defined as the maximum perpendicular distance between the interface of the myometrium and endometrium on the anterior and posterior walls of the uterine cavity, obtained from the largest sagittal section of the uterus.

SECONDARY OUTCOMES:
Vaginal bleeding volume | 14 days post-surgery
  Assessed by investigator-conducted follow-up interview at 14 days postoperatively. The postoperative vaginal bleeding volume is categorized as less, moderate, or more based on the subject's subjective perception, compared with her pre-operative menstrual flow volume.
Vaginal bleeding duration | 14 days post-surgery
  Assess the duration of vaginal bleeding after induced abortion surgery, measured in hours/days (recorded from the end of surgery until bleeding stops).
Time to menstrual resumption after abortion | Followed up and recorded within 60 days after induced abortion surgery (if no menstruation occurs by day 60, it will be recorded as "no resumption within 60 days").
  Time interval from the date of induced abortion surgery to the first day of spontaneous vaginal bleeding that meets the patient's usual menstrual flow volume and duration.
Changes in menstrual blood volume at first menstrual period post-abortion | Assessed at the end of the first menstrual period after abortion, with follow-up and recording completed within 60 days post-abortion.If no menstruation occurs by day 60, it will be recorded as "no resumption within 60 days".
  Compare the blood volume of the first menstrual period after abortion with the patient's pre-pregnancy usual menstrual blood volume (assessed via patient-reported sanitary product usage).

OTHER OUTCOMES:
Abnormality rate of blood, biochemical, and hormonal indicators | Pre-surgery: All 8 abovementioned indicators are tested and included in the abnormality rate calculation. 21 ± 2 days post-surgery: Only liver function tests, kidney function tests, estradiol and progesterone levels are tested.
  This outcome measures the proportion of participants with at least one abnormal indicator result. An indicator is defined as abnormal if its value falls outside the clinical normal reference range. The calculation formula is: (Number of participants with ≥1 abnormal result / Total eligible participants) × 100%. Included indicators cover routine blood tests, routine urine tests, coagulation function tests, routine vaginal discharge examination, liver function tests, kidney function tests, estradiol and progesterone levels (specific indicators tested differ by time frame).
Positive rate of bacterial culture on intrauterine stent surface | After stent removal at 21±2 days after surgery
  This outcome measure assesses intrauterine stent-related infection risk by culturing the patient's fluid samples from the stent surface. The specific method is to gently wipe the stent surface with a sterile swab to collect the patient's fluid. The "positive rate of bacterial culture on intrauterine stent surface" refers to the proportion of stents with positive bacterial culture results.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Dongcheng, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR